CLINICAL TRIAL: NCT00867932
Title: An Open-Label Multi-Center Study of Eculizumab in Children and Adolescents With a Diagnosis of Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Eculizumab Pharmacokinetics/Pharmacodynamics Study in Pediatric/Adolescent Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M07-005; 2009-010402-11 (EudraCT Number)
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Hemoglobinuria, Paroxysmal
Keywords: Alexion; Eculizumab; Paroxysmal Nocturnal Hemoglobinuria; PNH; Soliris
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Eculizumab (Experimental): Eculizumab was administered as an IV infusion for 12 weeks. All participants weighed more than 45 kg and received the following weight-based dosing regimen: induction/loading = 600 milligram (mg) weekly x 4; maintenance = 900 mg at Week 5; 900 mg every 2 weeks.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — 5 mg/mL solution in 5% Dextrose
  Other Names: Soliris®

SUMMARY:
The primary objective of this study was to evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) parameter estimates of eculizumab to confirm the dose regimens for pediatric and adolescent participants with PNH.

DETAILED DESCRIPTION:
This was an open-label, multi-center study of eculizumab administered to approximately 6 to 8 pediatric and adolescent participants aged 2 to 17 years with PNH. There were 3 periods in this study (screening, treatment, and post-treatment) with the treatment period having 2 dosing phases (induction and maintenance). If all screening criteria were met, the participant was eligible to enter the treatment period of the study after receiving Neisseria meningitidis (N. men), Streptococcus pneumoniae (S. pneumo), and Haemophilus influenzae (H. influ) vaccinations at least 14 days prior to first dose of study drug, or was vaccinated and received treatment with appropriate antibiotics until 14 days after the vaccinations. Participants received eculizumab intravenously (IV) based on their weight. Eculizumab was administered via an IV infusion at a rate of 5 to 10 milliliters (mL) per kilogram (kg) per hour (hr) (mL/kg/hr) for at least 25 minutes. The planned duration of treatment was 12 weeks with a 4-week induction phase and an 8-week maintenance phase. At the Investigator's and parents/legal guardian's discretion, participants who completed this study with eculizumab could continue treatment with commercially available eculizumab (Soliris®) and were followed in the Soliris® PNH Registry. Participants who stopped study participation before study completion or who did not continue with Soliris® treatment at the completion of the study were followed for 8 weeks and monitored for signs and symptoms of serious hemolysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 2 and 17 years of age;
* Diagnosed with PNH;
* Participants with ≥ 5% glycosylphosphatidylinositol-deficient red blood cells or granulocytes as confirmed by flow cytometry;
* Participants must have shown evidence of hemolytic anemia as documented by lactate dehydrogenase greater than the upper limit of normal or at least 1 transfusion in the past 2 years for anemia or anemia related symptoms;
* Written informed consent from a parent/guardian;
* Negative pregnancy test for females of child bearing potential at screening;
* Sexually active females must have documented a reliable and medically approved method of contraception;
* Participant must have been vaccinated against N. men, S. pneumo, and H. influ at least 14 days prior to study drug initiation or received antibiotics for 14 days after the vaccinations.

Exclusion Criteria:

* Prior eculizumab treatment;
* Presence or suspicion of active bacterial infection at baseline;
* Participation in another concurrent clinical study within at least 30 days prior to screening;
* History of meningococcal/pneumococcal/gonococcal disease;
* Pregnant, breast feeding, or intending to conceive during the study including the safety follow-up visits;
* Any other condition that could increase the participant's risk or confound the outcome of the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2009-10-02 (Actual); Primary Completion 2011-05-12 (Actual); Study Completion 2011-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orange, California
  - Pensacola, Florida
  - Memphis, Tennessee

REFERENCES:
- [Background] Reiss UM, Schwartz J, Sakamoto KM, Puthenveetil G, Ogawa M, Bedrosian CL, Ware RE. Efficacy and safety of eculizumab in children and adolescents with paroxysmal nocturnal hemoglobinuria. Pediatr Blood Cancer. 2014 Sep;61(9):1544-50. doi: 10.1002/pbc.25068. Epub 2014 Apr 29. PMID 24777716
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pubmed/24777716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period lasted from October 2009 to January 2011. Three sites in the United States of America enrolled a total of 7 participants with paroxysmal nocturnal hemoglobinuria (PNH).
Pre-assignment Details: Participants who completed this study could have continued treatment with commercially available eculizumab (Soliris®) and been followed in the Soliris® PNH Registry. Those who didn't complete the study or who didn't continue with Soliris® treatment after the study were followed for 8 weeks and monitored for signs and symptoms of serious hemolysis.
Groups:
- Eculizumab: Eculizumab was administered as an intravenous (IV) infusion for 12 weeks. All participants weighed more than 45 kilograms (kg) and received the following weight-based dosing regimen: induction/loading = 600 milligram (mg) weekly x 4; maintenance = 900 mg at Week (Wk) 5; 900 mg every 2 weeks (Q2W).
Period: Overall Study
Arm/Group | Eculizumab
Started | 7
Induction Phase | 7
Maintenance Phase | 7
Received at Least 1 Dose of Study Drug | 7
Intent-to-Treat (ITT) Population (Participants who received at least 1 dose of study drug.) | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: ITT Population: Participants who received at least 1 dose of study drug.
Groups:
- Eculizumab: Eculizumab was administered as an IV infusion for 12 weeks. All participants weighed more than 45 kg and received the following weight-based dosing regimen: induction/loading = 600 mg weekly x 4; maintenance = 900 mg at Wk 5; 900 mg Q2W.
Arm/Group | Eculizumab
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.01 (2.28)
Age, Customized [Count of Participants; unit: Participants]
  Children (2 to 11 years) | 1
  Adolescents (12 to 17 years) | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Peak And Trough Concentrations Of Eculizumab In Serum At Week 12
Description: Serum concentrations of eculizumab were measured by using a validated enzyme-linked immunosorbent assay (ELISA) method developed at Alexion Pharmaceuticals Bioanalytical Laboratory. The range of the analytical assay was 10 to 600 microgram per milliliter (μg/mL). Peak concentrations were not measured at the early termination (ET) visit.
Time Frame: Pre-infusion and 1 hour post-infusion at End of Treatment (EOT) (Day 84 [Week 12]) or ET
Population: ITT Population: Participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Eculizumab
Number analyzed (Participants) | 7
μg/mL
  Trough concentration | 192.5 [124.2 to 321.1]
  Peak concentration | 425.4 [220.5 to 566.1]

2. Secondary Outcome: Number Of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event (AE) not present prior to exposure to eculizumab or any event already present that worsened in either intensity or frequency following exposure to eculizumab. A serious TEAE was defined as any event that resulted in death, was immediately life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect. Related TEAEs were considered by investigators to be definitely, probably, or possibly related to administration of the study drug. Relationship is ordered as follows: unrelated, possibly related, probably related, or definitely related. TEAEs and TEAE severity were classified in accordance with the Medical Dictionary for Regulatory Activities (MedDRA) 13.0 dictionary. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: First dose of study drug (Day 0) to End of Follow-up (Week 20 [8 weeks after EOT])
Population: ITT Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 7
Participants
  Participants with at least 1 TEAE | 7
  Participants with any serious TEAE | 2
  Participants with any mild TEAE | 4
  Participants with any moderate TEAE | 1
  Participants with any severe TEAE | 2
  Participants with any unrelated TEAE | 2
  Participants with any possibly related TEAE | 3
  Participants with any probably related TEAE | 2
  Participants with any definitely related TEAE | 0

3. Secondary Outcome: Area Under The Curve (AUC) Of The Change From Baseline To Week 12 In Levels Of Lactate Dehydrogenase (LDH)
Description: The AUC of LDH was calculated by using the change of LDH from baseline values for each participant up to Week 12. For those participants with missing LDH values, the last observation carried forward method (LOCF) was used to impute missing values. Individual AUC values of LDH were summarized and tabulated.
Time Frame: Baseline, EOT (Day 84 [Week 12]) or ET
Population: ITT Population: Participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units * Days per Liter (U*Day/L)
Arm/Group | Eculizumab
Number analyzed (Participants) | 7
Units * Days per Liter (U*Day/L) | -60634 (72916)

4. Secondary Outcome: Concentration Of Plasma-free Hemoglobin At Baseline And Week 12
Description: Plasma-free hemoglobin was determined for each participant by using standard laboratory assays. The values of plasma-free hemoglobin were summarized by visit.
Time Frame: Baseline, EOT (Day 84 [Week 12]) or ET
Population: ITT Population: Participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg per deciliter (mg/dL)
Arm/Group | Eculizumab
Number analyzed (Participants) | 7
mg per deciliter (mg/dL)
  Baseline | 17.70 (19.091)
  Week 12 | 7.44 (3.145)

5. Secondary Outcome: Change From Baseline In LDH Levels
Description: Levels of LDH were determined by using standard laboratory assays. LDH values and the change of LDH from baseline were summarized by visit.
Time Frame: Baseline, Weeks 1 to 12 or ET
Population: ITT Population: Participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 7
U/L
  Baseline | 1020 (967)
  Change from baseline at Week 1 | -672 (837)
  Change from baseline at Week 2 | -763 (916)
  Change from baseline at Week 3 | -752 (934)
  Change from baseline at Week 4 | -761 (924)
  Change from baseline at Week 8 | -747 (904)
  Change from baseline at Week 12 | -771 (914)

ADVERSE EVENTS:
Time Frame: First dose of study drug (Day 0) to End of Follow-up (Week 20 [8 weeks after EOT])
Arm/Group | Eculizumab
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Eculizumab (N=7)
Anaemia (Blood and lymphatic system disorders) | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1/4 — Includes only female participants.
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/4 — Includes only female participants.
Acute sinusitis (Infections and infestations) | 1
Catheter site cellulitis (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Eculizumab (N=7)
Haemolysis (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Blood glucose increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 5
Chromaturia (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1/4 — Includes only female participants.
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/4 — Includes only female participants.
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes